CLINICAL TRIAL: NCT04357821
Title: Combinatorial Therapy With a Therapeutic Conserved Element DNA Vaccine, MVA Vaccine Boost, TLR9 Agonist and Broadly Neutralizing Antibodies: a Proof-of-concept Study Aimed at Inducing an HIV Remission
Brief Title: Combinatorial Therapy to Induce an HIV Remission
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); International AIDS Vaccine Initiative (Network); Ichor Medical Systems Incorporated (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Rockefeller University (Other); Mologen AG (Industry); GeoVax, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Deeks, Professor in Residence, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-26957
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination intervention arm (Experimental): All volunteers will receive the combination intervention outlined above.
  Interventions: Drug: Combination Intervention

INTERVENTIONS:
Drug: Combination Intervention — 1. IL-12 adjuvanted p24CE DNA prime (p24CE/IL-12) at Weeks 0 and 4
  2. IL-12 adjuvanted DNA boost (p24CE plus p55gag) at Week 12
  3. MVA/HIV62B (MVA62B) boost at Week 20
  4. single dose of two bNAbs (VRC07-523LS and 10-1074, which target CD4 binding site and V3 loop, respectively) at week 24 with a TLR9 agonist (lefitolimod) administered weekly between Weeks 24 and 33 (10 doses)
  5. ATI with single dose of VRC07 and 10-1074 at Week 34

SUMMARY:
Combination approaches will almost certainly be required to generate durable control of HIV in the absence of antiretroviral therapy (a "remission"). In this study, 20 individuals will receive a combination regimen administered during ART and then undergo an analytic treatment interruption (ATI).

DETAILED DESCRIPTION:
The investigators will perform a single arm study of twenty individuals with HIV infection on effective ART. All participants will receive a combination regimen administered during ART and then undergo an analytic treatment interruption. Our strategy has five stages

1. IL-12 adjuvanted p24CE DNA prime (p24CE/IL-12) at Weeks 0 and 4
2. IL-12 adjuvanted DNA boost (p24CE plus p55gag) at Week 12
3. MVA/HIV62B (MVA62B) boost at Week 20
4. single dose of two bNAbs (VRC07-523LS and 10-1074, which target CD4 binding site and V3 loop, respectively) at week 24 with a TLR9 agonist (lefitolimod) administered weekly between Weeks 24 and 33 (10 doses)
5. ATI with single dose of VRC07 and 10-1074 at Week 34

Follow-up off ART will occur through at least Week 46 (expected) and on or off ART (depending on outcome) through Week 86.

Should this approach work, viral load would be expected to rebound in all individuals a few weeks after the bNAb levels decrease to sub-therapeutic levels. This acute rebound would be followed by a new lower viral load set-point and perhaps a long-term remission.

ELIGIBILITY:
Key Inclusion Criteria

1. Willing and able to provide written informed consent.
2. Age ≤67 years at the time of enrollment for those who started treatment during early infection and <65 years for those who started treatment during chronic infection.
3. Documented HIV-1 infection.
4. On continuous antiretroviral therapy for at least 12 months without any interruptions of greater than 14 consecutive days within the last 1 year, and on a stable regimen that does not include an non-nucleoside reverse transcriptase inhibitor (NNRTI) for at least 4 weeks, without plans to modify ART during the study period.
5. Screening plasma HIV RNA levels below the level of quantification on all available determinations in past 24 months.
6. Screening CD4+ T-cell count ≥ 500 cells/mm3.

Key Exclusion Criteria

1. Subjects receiving a non-nucleoside reverse transcriptase inhibitor
2. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
3. High-level resistance to both 10-1074 and VRC-07 as defined using the PhenoSense Neutralizing Antibody Assay (Monogram Biosciences).
4. Any history of an HIV-associated malignancy, including Kaposi's sarcoma and any type of lymphoma, or virus-associated cancers.
5. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months.
6. CD4+ T cell nadir <350 cells/mm3 during the chronic phase of infection (beginning 6 months following the estimated infection date and confirmed on repeat testing).
7. Active hepatitis B (HBV) infection defined as positive HBV surface antigen test.

9. Active hepatitis C (HCV) infection. 10. Presence of significant abnormalities on electrocardiogram. 11. History of potential immune-mediated medical conditions. Individuals with isolated Raynaud's phenomenon or localized disease requiring topical therapy alone will not be excluded.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experience a new grade 3 or greater adverse event | Week 0 through 86
Proportion of participants achieving post-treatment control. | Week 34 through 86
  This will be defined as:
  1. Participants who fail to show any consistent rebound above 400 copies RNA/mL between Week 12 of the ATI (when bNAb levels wane) and Week 36 of the ATI
  2. Participants who exhibit a rebound and eventually achieve 24 weeks of virus control will be considered as having achieved post-treatment control

SECONDARY OUTCOMES:
Occurrence of any unsolicited adverse events for 28 days after administration of each study agent | Week 0 through 62
Occurrence of any serious adverse events, medically attended adverse event, and potentially immune-mediated medical condition from the time of administration of the first study injection through 12 months after administration of the final study injection | Week 0 through 86
Occurrence of two consecutive measurements HIV RNA >200 copies/mL using conventional assays | Week 34 to 86
Resumptions of antiretroviral therapy after treatment interruption and the events that trigger them | Week 34 to 86
Frequency of confirmed declines (two consecutive measurements) in CD4+ T cell counts (> 50%) | Week 34 to 86
Frequency of confirmed declines (two consecutive measurements) to below 350 cells/mm3 | Week 34 to 86
Proportion experiencing any clinically defined episode of acute retroviral syndrome | Week 34 to 86
Magnitude of T cell responses | Week 14
Breadth of T cell responses | Week 14
  The proportion of participants with at least one additional epitope response at week 14 (2 weeks after last vaccination) compared to their baseline response

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg San Francisco General Hospital, University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peluso MJ, Sandel DA, Deitchman AN, Kim SJ, Dalhuisen T, Tummala HP, Tiburcio R, Zemelko L, Borgo GM, Singh SS, Schwartz K, Deswal M, Williams MC, Hoh R, Shimoda M, Narpala S, Serebryannyy L, Khalili M, Vendrame E, SenGupta D, Whitmore LS, Tisoncik-Go J, Gale M Jr, Koup RA, Mullins JI, Felber BK, Pavlakis GN, Reeves JD, Petropoulos CJ, Glidden DV, Spitzer MH, Gama L, Caskey M, Nussenzweig MC, Chew KW, Henrich TJ, Yukl SA, Cohn LB, Deeks SG, Rutishauser RL. Correlates of HIV-1 control after combination immunotherapy. Nature. 2025 Dec 1. doi: 10.1038/s41586-025-09929-5. Online ahead of print. PMID 41326736